CLINICAL TRIAL: NCT03557580
Title: A Randomized, Open Label, Balanced, Single Dose, 3-way Crossover Bioequivalence Study of Two Isosorbide -5 -Mononitrate Extended -Release Tablets 40 mg and ISMO Retard 40 mg Under Fed Conditions in Healthy Subjects
Brief Title: A Bioequivalence Study of Isosorbide-5-Mononitrate Extended-Release Tablets Under Fed Conditions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-YK1-039-Y01
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Isosorbide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IS-5-MN R (Active Comparator): Isosorbide-5-mononitrate extended-release tablet, Single oral dose 40mg
  Interventions: Drug: IS-5-MN R
- IS-5-MN T1 (Experimental): Isosorbide-5-mononitrate extended-release tablet, Single oral dose 40mg
  Interventions: Drug: IS-5-MN T1
- IS-5-MN T2 (Experimental): Isosorbide-5-mononitrate extended-release tablet, Single oral dose 40mg
  Interventions: Drug: IS-5-MN T2

INTERVENTIONS:
Drug: IS-5-MN R — single orally dose under fed conditions on day 1 of treatment period 1 for group 1, on day 1 of treatment period 2 for group 2, on day 1 of treatment period 3 for group 3.
  Other Names: ISMO Retard; IS-5-MN
  Arms: IS-5-MN R
Drug: IS-5-MN T1 — single orally dose under fed conditions on day 1 of treatment period 2 for group 1, on day 1 of treatment period 3 for group 2, on day 1 of treatment period 1 for group 3.
  Other Names: IS-5-MN
  Arms: IS-5-MN T1
Drug: IS-5-MN T2 — single orally dose under fed conditions on day 1 of treatment period 3 for group 1, on day 1 of treatment period 1 for group 2, on day 1 of treatment period 2 for group 3.
  Other Names: IS-5-MN
  Arms: IS-5-MN T2

SUMMARY:
The purpose of this trial is to compare the pharmacokinetic characteristics of two isosorbide -5 -mononitrate extended -release tablets 40 mg of Qilu Pharmaceutical Co., Ltd and ISMO Retard (isosorbide -5 -mononitrate extended -release tablet) 40 mg, distributed by RIEMSER Pharma GmbH.

Primary endpoints are Cmax, AUC(0-t) and AUC(0-inf). Secondary endpoints are Tmax, t1/2 and λz.

DETAILED DESCRIPTION:
Objectives: Primary Objective: To compare the pharmacokinetic characteristics of two isosorbide -5 -mononitrate extended -release tablets 40 mg of Qilu Pharmaceutical Co., Ltd, China and ISMO Retard (isosorbide -5 -mononitrate extended -release tablet) 40 mg, distributed by RIEMSER Pharma GmbH. following a single oral dose administration in healthy Chinese subjects under fed condition.

Secondary Objective: To monitor the safety profile of the subjects exposed to the Investigational Medicinal Product.

Study Design: a randomized, open label, balanced, 3-way crossover, single dose study under fed conditions.12 subjects will be randomized to one of the 3 treatment sequences. Each treatment sequence will consist of 3 periods, separated by a washout period of at least 7 days. For sequence 1, first reference drug, then test formulation 1 and test formulation 2 will be administered. The order for sequence 2 is test formulation 2, reference drug and test formulation 1. The order for sequence 3 is test formulation 1, test formulation 2 and reference drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should read, sign, and date an Informed Consent Form under the premise of fully understanding of this study including risks and requirements; are unable to follow the rules of this study, prior to any study procedures;
* Healthy male or non-pregnant, non-lactating female of age between 18 to 50 years (both inclusive);
* Body weight ≥ 50 kg for male and 45 kg for female, body mass index (BMI) within 19.0-25.0 Kg/m2;
* Subject (including male subject) has no fertility plan within the future 3 months and take reliable contraceptive (physical);
* Subject must agree to use an acceptable method of birth control such as sexual abstinence or barrier method of contraception from screening until 3 months after last dose of study drug;
* Subject is considered reliable and capable of adhering to the protocol visit schedule or medication intake according to the judgment of the investigator.

Exclusion Criteria:

* Subject has allergic constitution or hypersensitivity to the active substance or to isosorbide dinitrate, or rare hereditary problems of galactose intolerance or fructose intolerance, the Lapp lactase deficiency, glucose - galactose malabsorption or sucrase - isomaltase insufficiency.
* Subject has dysphagia or any disorder that may interfere with drug absorption, distribution, metabolism, or excretion, e.g. gastrointestinal, liver, kidney conditions.
* Subject has alcoholism history or drank excessive alcohol within 6 months prior to the study (who drinking more than 21 units of alcohol per week, 1 unit = 360 mL beer (5%) = 45 mL spirit (40%) = 150 mL red-wine (12%)), positive test results for breath alcohol test at baseline, or cannot stop alcohol intake during study.
* Subject smoking more than 5 cigarettes/nicotine-containing products a day within 3 months prior to screening, or refusing to abstain from smoking or consumption of tobacco products during the study.
* Subject has significant change in diet or exercise habits within 3 months prior to screening.
* Subject has any food restrictions or intolerance.
* Subject has hospitalization history or surgery within 3 months prior to screening.
* Subject has made a blood donation or had a comparable blood loss (>400ml) within 3 months prior to screening.
* Subject has participated in another study of an investigational medication within the last 3 months, or taking any drugs known to have a well established toxic potential to major organs within 3 months prior to study administration.
* Subject with clinically significant blood, kidneys, endocrine, gastrointestinal, respiratory, cardiovascular, hepatic, psychiatric, immunological and neurological disease.
* Subject in cases of marked low blood pressure (BP ≤ 90 mmHg systolic), aortic/mitral valve stenosis, severe anaemia, glaucoma, or using a phosphodiesterase 5 inhibitor.
* Subject has history of drug abuse within the past 5 years, using any recreational drugs within 3 months prior to screening, or positive test results for urine drug scan.
* Female subject in lactation period, or has positive pregnancy test result, or had unprotected sexual intercourse within 14 days prior to first drug administration, or refusing to take non-pharmacological contraception (such as condoms, intrauterine devices, contraceptive rings, ligation, etc.).
* Subject with clinically significant positive test results for: HIV, Hepatitis B surface antigen, Hepatitis C antibody or treponema pallidum.
* Subject used any drugs known to induce or inhibit hepatic drug metabolism within 28 days prior to study administration.
* Subject has any prescription medication or over the counter within the 14 days prior to study administration.
* Subject using caffeine or any other beverages or foods that might affect drug absorption, metabolism or excretion, include coffee, tea, coke, chocolate, Animal viscera, dragon fruit, mango, grapefruit, grapefruit beverages or foods, etc. beginning 48 hours before each study medication administration through each study confinement period.
* Subject took any vitamins or herbal medicines (includes herbs in the diet) beginning 48 hours before each study medication administration through each study confinement period.
* Subject has any illness during the screening stage.
* Subject has history of blood phobia or belonephobia.
* Subject has any condition, according to investigator's best judgement, that prevents the subject to participate in the trial, or unable to adhere with restrictions detailed in the informed consent or protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose and 0.5, 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 24.0 36.0 and 48.0 hr post-dose
  Maximum plasma Capecitabine concentration
AUC0-t | Pre-dose and 0.5, 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 24.0 36.0 and 48.0 hr post-dose
  The area under the plasma concentration time curve from zero to the last measurable concentration.
AUC0-∞ | Pre-dose and 0.5, 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 24.0 36.0 and 48.0 hr post-dose
  The area under the plasma concentration time curve from zero to infinity.

SECONDARY OUTCOMES:
Tmax | Pre-dose and 0.5, 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 24.0 36.0 and 48.0 hr post-dose
  Time of the maximum measured plasma concentration
Kel | Pre-dose and 0.5, 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 24.0 36.0 and 48.0 hr post-dose
  The elimination rate constant associated with the terminal (log-linear) portion of the curve. Estimated by linear regression of time vs. log concentration.
t½ | Pre-dose and 0.5, 1.0, 2.0, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 24.0 36.0 and 48.0 hr post-dose
  The terminal elimination half-life calculated by 0.693/Kel.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingyuan People's Hospital, Qingyuan, China